CLINICAL TRIAL: NCT01611636
Title: Clinical Characteristics of Allergy, Autoimmune and Rheumatic Diseases: A Ten Year Retrospective Study
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chien-Sheng Wu, Chief, Division of Rheumatology, Far Eastern Memorial Hospital
Other Study IDs: 100165-E
Record Dates: First submitted 2012-05-26; First posted 2012-06-05 (Estimated); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Allergy; Autoimmune Diseases; Rheumatic Diseases
Keywords: allergy; autoimmune diseases; rheumatic diseases
MeSH Terms: conditions — Hypersensitivity; Autoimmune Diseases; Rheumatic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The incidence and prevalence of the allergic, autoimmune and rheumatic diseases are different all over the world. The relative impact of gene and environment on diseases can be revealed by studies from different populations. National Health Insurance database in Taiwan provides a wealth of epidemiology study, which can contribute to the understanding of these diseases. However, national health care database did not contain test results and clinical details. The database of the hospital records can provide complimentary clinical details. Via the comparison of databases of the National health Institutes and the investigators hospital, the investigators hope that the characteristics and outcomes of these patients can be better understood.

DETAILED DESCRIPTION:
The incidence and prevalence of the allergic, autoimmune and rheumatic diseases are different all over the world. The relative impact of gene and environment on diseases can be revealed by studies from different populations.

National Health Insurance database in Taiwan provides a wealth of epidemiology study, which can contribute to the understanding of these diseases. However, national health care database did not contain test results and clinical details. The database of the hospital records can provide complimentary clinical details. Via the comparison of databases of the National health Institutes and the investigators hospital, the investigators hope that the characteristics and outcomes of these patients can be better understood.

Briefly, epidemiology of target disease such as age, sex, incidence and prevalence will be derived from national database. Medical source utilization such as medication and surgery related to target diseases is also available in national database, providing material for cost analysis. These data can be compared with hospital database to ensure validity and reliability.

The investigators study is intended to provide epidemiology of target disease and cost analysis. Interaction between diseases will also be explored.

Target diseases Allergic diseases: Asthma(ICD9 493.x),Steven-Johnson syndrome and other erythroderma (ICD9 695.x)

Autoimmune diseases: Thyroid disease (ICD9 246.x), Addison disease (ICD9 255.x), type 1 diabetes mellitus (250.x1)

Rheumatic diseases: gout (ICD9 274.x), SLE (ICD9 710.0 ), RA (ICD9 714.0), AS and spondylitis (ICD9 720.0&720.x), Psoriasis and psoriatic arthritis (ICD9 696.0), scleroderma (ICD9 710.1), Sjogren's syndrome (ICD9 710.2), dermatomyositis (ICD9 710.3), polymyositis (ICD9 710.4), ANCA vasculitis (WG 446.4, MPA, CSS, PAN ICD9 446.0) or vasculitis 447.6, Behcet's disease(ICD9 136.1), Temporal arteritis(ICD9 446.5), Takayasu arteritis (ICD9 446.7), Henoch-Schonlein purpura (ICD9 287.0)

ELIGIBILITY:
Inclusion Criteria:

* subjects with ICD9 coding fulfilling study subjects

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: National Health Insurance Research Database Far Eastern Memorial Hospital clinical database
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Incidence of target diseases | Up to ten years
  Population at risk of target diseases in database will be assessed up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: ChienSheng Wu, Master, Principal Investigator — Chief, Department of Rheumatic disease
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No
No IPD sharing, only sharing by publication